CLINICAL TRIAL: NCT06129877
Title: CHAMP App Feeding Difficulties Repository
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Lori Erickson, Principal Investigator, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00002753
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Feeding and Eating Disorders of Childhood; Gastrostomy; Feeding Disorder of Infancy and Childhood
Keywords: mHealth; Software Platform; asynchronous remote monitoring
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CHAMP App — CHAMP App software platform will have been used in other research studies to be included in the Feeding difficulties repository

SUMMARY:
This repository will consist of home monitoring data, videos, and images of patients with feeding difficulties for asynchronous remote patient monitoring of manually entered data sent by parents to the healthcare team using the CHAMP App for children with feeding difficulties. This information will be collected under a research protocol and this repository is for future research applications.

DETAILED DESCRIPTION:
Around 25% of children are reported to have some degree of feeding issues of whom 3-10% have more severe feeding disorders1. Many of these feeding issues and difficulties can also lead to a need for supplemental nutrition in a child's diet due to the impact on growth. Those requiring supplemental nutrition may find themselves having to be fed using tube feedings (TF), which carries its own set of obstacles and factors to consider. While feeding problems have been estimated to occur in 25%-35% of children observed as exhibiting normal growth, that number may spike to 85% in those with GI-related growth disorders2. This highlights the need to ensure treatment plans and programs are in place to assist this patient population.

At Children's Mercy Hospital, GI specialists care for children who have a variety of conditions, caring for the whole child and addressing physical, mental, emotional, and social aspects. By using a combined approach, and promoting research that seeks to improve care, significant improvements in children's health have been reported. One specialty this has been evident in at Children's Mercy is the cardiac patient population. There have been improvements in growth, feedings, and timeliness of interventions seen with the use of CHAMP® App in the single ventricle population (a statistically significant difference in the frequency of growth failure, with no patients having growth failure during CHAMP use)3-4. By harnessing the experience and knowledge gained through the CHAMP® App research study, there is a great potential for children suffering from GI conditions to also benefit from this form of remote patient management and monitoring, especially when it comes to treating children with supplemental nutrition needs. There are no known Gastroenterology- Feeding mobile health software platforms with a dedicated research repository in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolling in this research repository must also be enrolled in an applicable study (STUDY00002775, STUDY00003221) wherein they have consented to use CHAMP App
* Parent-Legally authorized representative can read one of the eleven languages that the CHAMP App is available in.

Exclusion Criteria:

• All patients and parents/Legally authorized representative not meeting the above specified criteria

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with feeding difficulties and/or malnutrition
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Feeding difficulty management | 12 months
  Percent of patients eating all calories by mouth at the end of asynchronous remote monitoring period for feeding management

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Director, Remote Health Solutions Children's Mercy
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided